CLINICAL TRIAL: NCT01745055
Title: A Phase 1, Open Label Study Of The Pharmacokinetics Of Multiple Doses Of Oral CP-690,550 And Single Doses Of Oral Methotrexate In Rheumatoid Arthritis Subjects
Brief Title: Co-Administration Of Methotrexate And CP-690,550
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921013
Record Dates: First submitted 2012-12-04; First posted 2012-12-07 (Estimated); Results first posted 2012-12-07 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Pharmacokinetics; oral JAK inhibitor; methotrexate (MTX); rheumatoid arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-690,550 (tofacitinib) 30 mg q12h (Experimental): Individual dose of methotrexate with the addition of CP-690,550 30 mg q12h
  Interventions: Drug: CP-690,550 (tofacitinib); Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: CP-690,550 (tofacitinib) — CP-690,550 30 mg q12h for 5 days
Drug: Methotrexate (MTX) — individual dose of methotrexate (stably dosed)

SUMMARY:
This study was designed to estimate the effects of methotrexate (MTX) on the pharmacokinetics (PK) of CP-690,550 when administered to subjects with rheumatoid arthritis (RA), to estimate the effects of CP-690,550 on the PK of MTX and to evaluate the short-term safety and tolerability of co-administration of CP-690,550 and MTX.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with moderate to severe RA (Rheumatoid Arthritis)
* Diagnosis of RA based on the American College of Rheumatology 1987 revised criteria.
* Treatment with an oral stable weekly dose of Methotrexate (MTX) (15-25 mg/week, administered as a single dose [SD]) for a minimum of 4 doses (4 weeks)

Exclusion Criteria:

* Blood dyscrasias including confirmed: Hemoglobin <9 g/dL or Hematocrit <30%; White blood cell count <3.0 x 109/L; Absolute neutrophil count <1.2 x 109/L; Platelet count <100 x 109/L
* Evidence or history of clinically significant infections within the past 6 months (eg, those requiring hospitalization, requiring parenteral antimicrobial therapy, or those with recurrent oral or genital herpes, recurrent herpes zoster, or any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the trial.
* Total bilirubin, AST (aspartate aminotransferase) or ALT (alanine aminotransferase) more than 1.2 times the upper limit of normal at the Screening visit, or a history of clinically significant elevated liver function tests (LFTs) while on current MTX dose or chronic liver disease, recent or active hepatitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Miramar, Florida
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921013&StudyName=Co-Adminstration%20Of%20Methotrexate%20And%20CP-690%2C550

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate + CP-690,550: Single oral dose of methotrexate (MTX) on Day 1 (15-25 milligram [mg], as per local prescribing practice); followed by CP-690,500 30 mg tablet orally every twelve hours from Day 3 to Day 6; followed by single oral dose of MTX (15-25 mg, as per local prescribing practice) and single oral dose of CP-690,500 30 mg tablet orally, on Day 7.
Period: Overall Study
Arm/Group | Methotrexate + CP-690,550
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methotrexate + CP-690,550
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to 12 Hours [AUC (0-12)] for CP-690,550
Description: AUC (0-12)= area under the plasma concentration time-curve from time zero (pre-dose) to 12 hours (0-12).
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8 and 12 hours post-dose on Day 6 and Day 7
Population: The pharmacokinetic (PK) analysis population included all enrolled participants with PK parameters of interest for at least 1 period of fixed sequence.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- CP-690,500: CP-690,500 30 mg tablet orally every twelve hours from Day 3 to Day 6.
- Methotrexate + CP-690,500: Single oral dose of MTX (15-25 mg, as per local prescribing practice) and single oral dose of CP-690,500 30 mg tablet orally, on Day 7.
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
nanogram*hour/milliliter (ng*hr/mL) | 1370 (423) | 1410 (425)
Statistical Analysis 1: Comparison: CP-690,500 vs Methotrexate + CP-690,500; Natural log transformed, AUC (0-12) of CP-690,550 was analyzed using mixed effect model with treatment as fixed effects and participant as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 103.06, 90% CI 2-sided [99.00 to 107.29]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for CP-690,550
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8 and 12 hours post-dose on Day 6 and Day 7
Population: The PK analysis population included all enrolled participants with PK parameters of interest for at least 1 period of fixed sequence.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
ng/mL | 375 (91.6) | 384 (84.8)
Statistical Analysis 1: Comparison: CP-690,500 vs Methotrexate + CP-690,500; Natural log transformed, Cmax of CP-690,550 was analyzed using mixed effect model with treatment as fixed effects and participant as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 102.71, 90% CI 2-sided [93.79 to 112.47]

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Methotrexate (MTX)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours post-dose on Day 1 and Day 7
Population: PK analysis population included all enrolled participants with PK parameters of interest for at least 1 period of fixed sequence.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Methotrexate: Single oral dose of MTX on Day 1 (15-25 milligram [mg], as per local prescribing practice).
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 1850 (685) | 1720 (753)
Statistical Analysis 1: Comparison: Methotrexate vs Methotrexate + CP-690,500; Natural log transformed, AUClast of MTX was analyzed using mixed effect model with treatment as fixed effects and participant as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 89.53, 90% CI 2-sided [77.38 to 103.57]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Methotrexate (MTX)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24 and 48 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Methotrexate: Single oral dose of methotrexate (MTX) on Day 1 (15-25 milligram [mg], as per local prescribing practice).
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
ng/mL | 478 (106) | 433 (175)
Statistical Analysis 1: Comparison: Methotrexate vs Methotrexate + CP-690,500; Natural log transformed, Cmax of MTX was analyzed using mixed effect model with treatment as fixed effects and participant as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 87.25, 90% CI 2-sided [76.03 to 100.12]

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for CP-690,550
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8 and 12 hours post-dose on Day 6 and Day 7
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
hour | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 1.00]

6. Secondary Outcome: Plasma Decay Half-Life (t1/2) for CP-690,550
Description: Plasma decay half-life is the time measured for the plasma concentration of CP-690,550 to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8 and 12 hours post-dose on Day 6 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
hour | 2.64 (0.356) | 3.12 (0.74)

7. Secondary Outcome: Apparent Oral Clearance (CL/F) for CP-690,550
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8 and 12 hours post-dose on Day 6 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
mL/hr | 23200 (8380) | 23511 (8784)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Methotrexate (MTX)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 ,12, 24 and 48 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
hour | 1.00 [0.50 to 1.50] | 1.25 [0.50 to 2.00]

9. Secondary Outcome: Plasma Decay Half-Life (t1/2) for Methotrexate (MTX)
Description: Plasma decay half-life is the time measured for the plasma concentration of MTX to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 , 12, 24 and 48 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
hour | 2.87 (0.962) | 3.36 (1.13)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) for Methotrexate (MTX)
Description: as for outcome 7
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 , 12, 24 and 48 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
mL/hr | 9890 (3370) | 11500 (5430)

11. Secondary Outcome: Total Amount of Unchanged Drug Excreted in the Urine From Time Zero to 12 Hours (Ae[0-12]) for CP-690,550
Time Frame: 0 (pre-dose) through 12 hours post-dose on Day 6 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
milligram | 6.65 (2.26) | 6.58 (2.34)

12. Secondary Outcome: Renal Clearance (CL R) for CP-690,550
Time Frame: 0 (pre-dose) through 24 hours post-dose on Day 6 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: litre/hour (L/hr)
Arm/Group | CP-690,500 | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
litre/hour (L/hr) | 5490 (2890) | 5240 (2630)

13. Secondary Outcome: Total Amount of Unchanged Drug Excreted in the Urine From Time Zero to 24 Hours (Ae[0-24]) for Methotrexate (MTX)
Time Frame: 0 (pre-dose) through 24 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
milligram | 18.1 (9.31) | 13.2 (4.38)

14. Secondary Outcome: Renal Clearance (CL R) for Methotrexate (MTX)
Time Frame: 0 (pre-dose) through 24 hours post-dose on Day 1 and Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Methotrexate | Methotrexate + CP-690,500
Number analyzed (Participants) | 12 | 12
L/hr | 10.2 (4.56) | 8.95 (4.64)

ADVERSE EVENTS:
Groups:
- Methotrexate: Single oral dose of MTX on Day 1 (15-25 mg), as per local prescribing practice.
Arm/Group | Methotrexate | CP-690,500 | Methotrexate + CP-690,500
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 6/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=12) | CP-690,500 (N=12) | Methotrexate + CP-690,500 (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0
Migrane (Nervous system disorders) | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Results were summarized for Ae(0-12) instead of planned Ae(0-24), as CP-690,550 was administered every 12 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.